CLINICAL TRIAL: NCT06588504
Title: A Phase 3, Randomised, Open-label, Cross-over Study to Confirm the Clinical Efficacy and Safety of Dasiglucagon Versus Glucagon for the Treatment of Severe Hypoglycaemia in Asian Adults With Type 1 Diabetes (T1D) Including an Investigation of Dasiglucagon in a Japanese Adolescent Cohort
Brief Title: Research Study in Japan to Compare Dasiglucagon With Glucagon in Treating Very Low Levels of Blood Sugar in Asian Adults With Type 1 Diabetes and Testing of Dasiglucagon for the Same Condition in Japanese Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9515-7675; U1111-1300-1855 (Other: World Health Organization (WHO)); jRCT2071240050 (Registry Identifier: Japan Registry for Clinical Trials (jRCT))
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dasiglucagon; Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Adult Cohort: Dasiglucagon then Glucagon (Experimental): Participants will receive a single subcutaneous (s.c.) injection of dasiglucagon in first dosing visit then a single intra-mascular (i.m.) injection of glucagon in next dosing visit.
  Interventions: Drug: Dasiglucagon
- Adult Cohort: Glucagon then Dasiglucagon (Experimental): Participants will receive a single i.m. injection of glucagon in first dosing visit then a single s.c. injection of dasiglucagon in next dosing visit.
  Interventions: Drug: Dasiglucagon; Drug: Glucagon
- Adolescent Cohort: Dasiglucagon (Experimental): Participants will receive a single s.c. injection of dasiglucagon.
  Interventions: Drug: Dasiglucagon

INTERVENTIONS:
Drug: Dasiglucagon — Participants will receive s.c. injection of dasiglucagon.
Drug: Glucagon — Participants will receive i.m. injection of glucagon.
  Arms: Adult Cohort: Glucagon then Dasiglucagon

SUMMARY:
This study will be looking to confirm the effect of dasiglucagon when compared with glucagon for treating very low sugar levels in Asian adults with T1D and the effect of dasiglucagon in Japanese adolescents with T1D. This study wants to demonstrate that dasiglucagon can raise low blood sugar levels just as well as glucagon. Participants will get dasiglucagon and glucagon. In which treatment order participants get study medicines (dasiglucagon and glucagon) is decided by chance. Dasiglucagon is a new medicine, but doctors can prescribe it in the US as it is approved there. Doctors can prescribe glucagon in multiple countries including Japan as an approved medicine. The study will last for about 17 weeks. Participant cannot be in the study if the study doctor thinks that there are risks for participants health. Women cannot take part if pregnant, breast-feeding, plan to get pregnant, during the study period, or not using adequate contraceptive methods. For man: if participant have sex, participant and his partner must use an adequate birth control method during the study.

ELIGIBILITY:
Inclusion Criteria:

* For Adults: Asian male or female; For Adolescents: Japanese male or female.
* Age at the time of signing the informed consent:

For Adults: Age 18-75 years (both inclusive):

For Adolescents: Age 12-15 years (both inclusive).

* Diagnosed with T1D greater than (>)1 year before screening.
* Glycated haemoglobin (HbA1c) less than (<)10.0 percentage (%) (86 millimoles per mole [mmol/mol]) as assessed by subcontracted laboratory by the site on the day of screening.
* For adults: BMI between 18.5 and 29.9 kilogram per meter square (kg/m2) (both inclusive).

For adolescents: Body weight greater than or equal to (≥) 33.4 kilograms (kg).

* Treated with stable insulin treatment (based on the investigator's discretion preferably no more than a 10-unit daily variation in total daily insulin dose) 30 days prior to screening.
* For Japanese participants: Japanese passport or equivalent For non-Japanese participants: Asian (non- Japanese passport or equivalent).

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products (glucagon or its derivatives).
* Exposure to an investigational medicinal product (IMP) within 30 days or 5 times the half-life of the IMP (if known), whichever is longest before screening.
* Severe hypoglycaemia in the last month prior to screening.
* Hospitalisation for diabetic ketoacidosis (DKA) in the last month prior to screening.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological conditions (except conditions associated with diabetes mellitus).
* History of epilepsy or seizure disorder.
* Known presence or history of pheochromocytoma (i.e., adrenal gland tumour) or insulinoma (i.e., insulin-secreting pancreas tumour).
* Clinically significant abnormal electrocardiogram (ECG) at screening as evaluated by investigator.
* Any disorder, unwillingness or inability which in the investigator's opinion, might jeopardise the participant's safety or compliance with the protocol.

As declared by the participant or in the medical records.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Adults cohort: Time to plasma glucose (PG) recovery, where PG recovery is defined as the first increase in PG of greater than or equal to (>=) 20 milligrams per decilitre (mg/dL) (1.1 millimoles per litre [mmol/L]) from baseline | From 0 to 90 minutes after investigational medicinal product (IMP) injection
  Measured in minutes.

SECONDARY OUTCOMES:
Adolescent cohort: Time to PG recovery, where PG recovery is defined as the first increase in PG of >=20 mg/dL (1.1 mmol/L) from baseline | From 0 to 90 minutes after IMP injection
  Measured in minutes.
PG recovery within 30 minutes after IMP injection (yes/no) | From 0 to 30 minutes after IMP injection
  Measured in count of participant.
PG recovery within 20 minutes after IMP injection (yes/no) | From 0 to 20 minutes after IMP injection
  Measured in count of participant.
PG recovery within 15 minutes after IMP injection (yes/no) | From 0 to 15 minutes after IMP injection
  Measured in count of participant.
PG change from baseline at 15 minutes after IMP injection | From 0 to 15 minutes after IMP injection
  Measured in milligrams per deciliter (mg/dL).
PG change from baseline at 20 minutes after IMP injection | From 0 to 20 minutes after IMP injection
  Measured in mg/dL.
Area under the plasma dasiglucagon concentration time curve after IMP injection | On Day 1 after injection
  Measured in hour*picomoles per liter (h*pmol/L).
Maximum observed plasma (Cmax) dasiglucagon concentration | From 0 to 5 hours after IMP injection
  Measured in pmol/L.
Number of adverse events (AEs) | From IMP injection (visit 2 day 1 and visit 3 day 1) until 28 days after IMP injection
  Measured in number of events.
Number of hypoglycaemic episodes | From IMP injection (visit 2 day 1 and visit 3 day 1) until 12 hours after IMP injection
  Measured in number of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Hakata Clinic, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com